CLINICAL TRIAL: NCT06362824
Title: De Pie y a Movernos Study: Promoting Physical Activity in Older Hispanic/Latino(a) Adults
Brief Title: Promoting Physical Activity in Older Hispanic/Latino(a) Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2094138
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Sedentary Behavior; Physical Inactivity; Alzheimer Disease, Protection Against
MeSH Terms: conditions — Sedentary Behavior; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- De Pie Intervention (Experimental): The De Pie intervention program receives a sedentary behavior reduction and physical activity promotion intervention centered on two steps: Step 1) reduce sitting time and move more throughout the day; Step 2) if cleared by a safety assessment and blood pressure check, participants can work towards adding structured bouts of exercise into their day.
  Interventions: Behavioral: De Pie Intervention
- HALT-AD Active Comparison Group (Active Comparator): Those randomized to HALT-AD (Healthy Actions and Lifestyles to Avoid Dementia) will receive one phone call to introduce them to preventing cognitive decline through various lifestyle behaviors (e.g. stress reduction, healthy diet, healthy sleep) other than physical activity. They will be encouraged by the Health Coach upon randomization to complete one module approximately every week (there are 10 modules in total).
  Interventions: Other: Active Comparison Group: Healthy Actions And Lifestyles To Avoid Dementia (HALT-AD)

INTERVENTIONS:
Behavioral: De Pie Intervention — Participants are guided by a health coach trained in motivational interviewing through 6 biweekly phone sessions. Each session involves reviewing goals and problem-solving barriers from the prior 2 weeks experience; covering a topic related to Step 1 goals (or Step 2 goals if they pass the safety assessment) such as how to enjoy movement, social support, and using your surroundings; and setting goals and an action plan for the following two weeks.
  Arms: De Pie Intervention
Other: Active Comparison Group: Healthy Actions And Lifestyles To Avoid Dementia (HALT-AD) — Those in the active comparison program will receive no additional health coaching sessions. They will work through the HALT-AD content at their own pace, setting goals in the online platform as they go.
  Arms: HALT-AD Active Comparison Group

SUMMARY:
In this randomized controlled trial, study staff will randomize 130 Hispanic/Latino adults without dementia and over age 55 from Southern California and from Kaiser Permanente Washington (State) to either the culturally adapted De Pie physical activity intervention or an active comparison program focusing on general brain health topics. The purpose of this study is to determine if 12 weeks of the culturally adapted and fully remote De Pie y a Movernos intervention improves self-efficacy, habit strength, social support, and enjoyment for physical activity (PA), thus promoting adherence to moderate-intensity physical activity (MIPA) guidelines (150 minutes/week).

DETAILED DESCRIPTION:
Building on the cultural adaptation of our preliminary R61 De Pie pilot study, study staff will randomize 130 Hispanic/Latino adults without dementia and over age 55 from Southern California and from Kaiser Permanente Washington to either the culturally adapted De Pie physical activity intervention or an active comparison program, Healthy Actions and Lifestyles to Avoid Dementia (HALT-AD), focusing on general brain health topics. The investigators will determine if De Pie improves physical activity (Aim 1) and psychosocial mediators (self-efficacy, habit strength, social support, and enjoyment for physical activity, [PA]), thus promoting adherence to moderate-intensity physical activity (MIPA) guidelines (150 minutes/week; Aim 2). The intervention period lasts 12 weeks.

The investigators target middle-aged and older Hispanic/Latino adults that are under-studied and have a higher risk of Alzheimer's disease and related dementias (ADRD), compared to non-Hispanic White older adults. Study staff employ a community engaged and collaborative approach to culturally adaptive the intervention framework and a staircase intervention approach designed to build self-efficacy, PA habit strength, social support, and PA enjoyment. Results will inform culturally adapted, theory-based approaches to prevent ADRD in the Hispanic/Latino community.

ELIGIBILITY:
Inclusion Criteria:

* be 55-89 and self-identify as Hispanic/Latino(a)
* able to participate for up to 20 weeks in the study
* willing to be randomized to the intervention or active comparison program
* willing to follow study procedures depending on program assignment
* available M-F for study phone calls between 8am-5pm
* able to walk one block unassisted,
* able to speak and can read Spanish or English,
* have a smartphone (85% of the Hispanic/Latino(a) population has a smartphone)
* willing to wear an ActiGraph for up to 2 weeks, twice during the course of the study
* willing to complete study questionnaires via weblink, paper, or phone call
* have an email address and be willing to share it with the team
* have a US mailing address where they receive mail regularly (confirmed in pre-screen)

Exclusion criteria are as follows:

* score less than or equal to 4 on the Six-Item Screener (Callahan et al., 2002)
* unable to hear phone conversation, even with a hearing aid
* planned surgeries or travel that would interfere with participation
* had a fall in the last year that resulted in hospitalization
* had a cancer diagnosis that requires treatment in the past year (other than skin cancer)
* had a diagnosis of heart attack or irregular heart beat (arrythmia) in the past year
* been advised recently by their doctor to avoid physical activity
* does not want to share cognitive health information collected during the study with researchers at UCSD
* unwilling to share their email address
* unwilling to obtain an email address if they do not already have one
* currently participating in another institution's physical activity study

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Moderate Intensity Physical Activity (MIPA) minutes/day | Baseline to 12 weeks
  Time (minutes) spent being physically active during waking hours will be measured objectively by the ActiGraph worn for one week at Baseline and again after 12 weeks

SECONDARY OUTCOMES:
Meet MIPA guidelines of 150 minutes physical activity per week | Baseline to 12 weeks
  Time (minutes) spent being physical active during waking hours will be measured objectively by the ActiGraph worn for one week at Baseline and again after 12 weeks
Average daily sedentary time | Baseline to 12 weeks
  mins/day; ≤18 counts per 15s will be measured objectively by the ActiGraph worn for one week at baseline and again after 12 weeks.
Average daily light intensity physical activity (LPA) | Baseline to 12 weeks
  mins/day; 19-518 counts per 15s will be measured objectively by the ActiGraph worn for one week at Baseline and again after 12 weeks
Average steps/day | Baseline to 12 weeks
  Change in daily steps will be measured objectively by the ActiGraph worn for one week at Baseline and again after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dori E Rosenberg, PhD, MPH, Principal Investigator — Kaiser Permanente; Zvinka Z Zlatar, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Kaiser Permanente Washington, Seattle, Washington